CLINICAL TRIAL: NCT07347639
Title: SOCAV: a Nurse-led Support Programme for Self-direction in People With Dementia in Dutch Home Care, Involving Informal Caregivers - a Feasibility Study With Process Evaluation
Brief Title: SOCAV: a Nurse-led Support Programme for Self-direction in People With Dementia
Acronym: SOCAV-program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MEC A-N 2019-5689
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Dementia Caregivers
Keywords: SOCAV; Caregivers; Primary care; Nursing care; Person-centered care; Feasibility study
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This is a single-group, non-randomized feasibility study with a longitudinal pre-post evaluation and embedded process evaluation. All enrolled participants received the SOCAV-Home Care program (there was no control or comparison arm). The intervention was delivered at the level of the home-care team/nurses (training plus ongoing reflective coaching over approximately 6-9 months), with dyad-level components for the person with dementia and informal caregiver (a series of collaborative home meetings over approximately 3-6 months). Outcomes were assessed repeatedly over time (baseline and follow-up time points during the intervention period) to explore feasibility and signals of potential benefit rather than to test efficacy.
Masking Description: Not applicable. This was a single-arm feasibility study and no additional parties were formally masked/blinded; participants (people with dementia and informal caregivers), nurses, peer coaches, and the research team were aware of the intervention. Interviewers were independent/unknown to participants, but they were not blinded to intervention exposure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOCAV-Home Care intervention arm (Other): Single-arm study: all participants received SOCAV-Home Care, where home-care nurses were trained and coached to support autonomy in daily decisions, and the person with dementia and caregiver had several home sessions to set goals and agree on practical strategies to maintain choice and independence.
  Interventions: Behavioral: SOCAV-Home Care (self-directed care support for home-dwelling people with dementia)

INTERVENTIONS:
Behavioral: SOCAV-Home Care (self-directed care support for home-dwelling people with dementia) — SOCAV-Home Care is distinct because it targets "self-direction" in everyday home-care situations by combining (1) structured nurse training in person-centered communication (based on Community Occupational Therapy in Dementia principles), (2) longitudinal Kalorama reflective coaching with reflective diaries to change routine nursing behavior over months, and (3) repeated triadic home sessions (person with dementia + informal caregiver + nurse, sometimes with a peer coach) focused on mapping preferences, setting shared goals, and testing practical autonomy-supporting strategies in the home context. It is implemented by trained peer coaches within home-care teams rather than as a stand-alone therapy delivered only to patients.
  Other Names: SOCAV program; SOCAV home care

SUMMARY:
In this study, we tested whether a support program could help people living at home with dementia keep making their own everyday choices for as long as possible, with help from a family caregiver and a home-care nurse. Nurses received training and coaching to better focus on what the person still wants and can do, and to avoid taking over tasks too quickly. The program also included home conversations with the person with dementia and their caregiver to agree on what matters most and how to support that in daily life. In total, 12 people with dementia, 14 caregivers, and 33 nurses took part. Most participants felt the program was helpful and said it increased attention to personal choice and small day-to-day decisions. However, it also took time and was sometimes hard to schedule, and some people dropped out. The questionnaires did not show clear improvements in things like quality of life, but there were signs that some behavior problems (such as restlessness or difficult situations) became less frequent for some participants.

ELIGIBILITY:
Inclusion Criteria:

* People with dementia were eligible if they had mild to moderate dementia (diagnosed by a general practitioner or geriatrician), lived at home, and received care from a home-care team.
* Informal caregivers were eligible if they provided care at least twice per week, either as a co-residing primary caregiver or as a regularly visiting secondary caregiver.
* Nurses were eligible if they worked in home care, supported people with dementia, and were employed by the regional care organization.

Exclusion Criteria:

* People with dementia were excluded if they had a Geriatric Depression Scale (GDS) score >6;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | The COPM was administered at baseline and 5 months in the development phase, and in the feasibility phase at baseline, 4 months (midpoint), and 9 months (endpoint).
  The Canadian Occupational Performance Measure (COPM) (Dutch version) is a tool to assess change in performance of meaningful daily activities and satisfaction with that performance, each rated on a 1-10 scale (1 = not able/not satisfied at all; 10 = fully able/fully satisfied), based on input from the person with dementia, the informal caregiver, and the home-care nurse.
  Main Manuscript
Canadian Occupational Performance Measure | The COPM was administered at baseline and 5 months in the development phase, and in the feasibility phase at baseline, 4 months (midpoint), and 9 months (endpoint).
  The Canadian Occupational Performance Measure (COPM) (Dutch version) is a tool to assess change in performance of meaningful daily activities and satisfaction with that performance, each rated on a 1-10 scale (1 = not able/not satisfied at all; 10 = fully able/fully satisfied), based on input from the person with dementia, the informal caregiver, and the home-care nurse.

SECONDARY OUTCOMES:
The Dementia Quality of Life (DQoL) | The DQoL was collected as a primary outcome at baseline, 4 months (midpoint), and 9 months (endpoint) in the feasibility phase (and at baseline and 5 months in the development phase).
  The Dementia Quality of Life (DQoL) is a 29-item, dementia-specific quality-of-life measure that is administered as an interview with the person living with dementia and is intended for people with mild to moderate dementia. It captures the person's own view of their quality of life across key concepts including self-esteem, positive affect/humor, absence of negative affect, feelings of belonging, and sense of aesthetics.
Centre for Epidemiologic Studies Depression Scale (CES-D), | In the feasibility phase, the CES-D was assessed at baseline, 4 months, and 9 months (and at baseline and 5 months in the development phase).
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a brief questionnaire used to assess depressive symptoms (more symptoms = higher score). In this study it was used with informal caregivers.

OTHER OUTCOMES:
Reflective coaching diaries | Nurses completed these continuously throughout the reflective coaching period, starting after the training and continuing until the end of the program, i.e., over approximately 6-9 months (from baseline through the feasibility endpoint).
  Reflective coaching diaries (nurses): qualitative assessment of feasibility/implementation and changes in attitudes/behaviors, analyzed with constant comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Avoord, Etten-Leur, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Due to confidentiality and the risk of re-identification in this small sample, we will not publicly share qualitative interview/focus group transcripts, reflective diaries, or other qualitative materials. However, de-identified individual-participant quantitative data underlying the published results (e.g., COPM, DQoL, CES-D and other questionnaire outcomes), together with a data dictionary/codebook and the analytic code used for the published analyses, are available upon reasonable request.
Supporting Information: ICF, CSR, Analytic Code
Time Frame: Starting at publication of the primary results; ending 5 years after publication.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to de-identified individual-participant quantitative data underlying the published results, together with a data dictionary/codebook and the analytic code used for the published analyses. Requests will be reviewed by the study team and, if approved, data will be shared under a signed data use agreement (and ethics approval if required), via secure file transfer or a controlled-access repository.
URL: http://radboudumc.nl

REFERENCES:
- [Background] Corporaal, Sharissa & Huijbregts, Ralf & Graff, Maud. (2019). SOCAV: persoonsgerichte zorg bij dementie. Bijblijven. 35. 40-45. 10.1007/s12414-019-0020-z. https://www.researchgate.net/publication/331740573_SOCAV_persoonsgerichte_zorg_bij_dementie
- See also: SOCAV helps people with dementia keep autonomy and meaningful daily activities. It trains family and professional caregivers to reflect, optimize, compensate and teach skills, supporting clients to live at home longer with enjoyment and dignity. — https://www.dementievriendelijk.nl/projecten/zorgconcept-socav-in-de-thuissituatie